CLINICAL TRIAL: NCT06867588
Title: The Added-value of PSMA PET in Detecting Clinically Significant Prostate Cancer Lesions in Patients Undergoing MRI-targeted Biopsy. (PANDORA): a Prospective, Paired Diagnostic Study
Brief Title: The Added-value of PSMA PET in Detecting Clinically Significant Prostate Cancer Lesions in Patients Undergoing MRI-targeted Biopsy. (PANDORA)
Acronym: PANDORA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJBPANDORA
Record Dates: First submitted 2025-02-25; First posted 2025-03-10 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-02

CONDITIONS: Multiparametric MRI; Lesion PI-RADS 3
Keywords: PSMA PET; MRI-targeted biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with at least one lesion PI-RADS 3 (Other)
  Interventions: Diagnostic Test: PSMA PET

INTERVENTIONS:
Diagnostic Test: PSMA PET — patients included in the study will perfom a PSMA PET

SUMMARY:
Prostate Specific Membrane Antigen (PSMA) positron emission tomography/computed tomography (PET/CT), an imaging modality focusing on a protein overexpressed by prostate cancer cells, has revolutionised the staging of both newly diagnosed and biochemically recurrent prostate cancer with better performance when compared to conventional imaging. Indeed, several studies have shown that PSMA PET/CT outperformed choline PET/CT with better detection rate of metastatic disease, particularly in the setting of disease recurrence after therapy even at (very) low PSA level. Moreover, the proPSMA trial reported that PSMA PET/CT had 27% greater accuracy than that of CT and bone scanning when staging patients with high-risk localised prostate cancer. More recently, availability of integrated PET/MRI scanners offers the opportunity for higher accuracy imaging and promising diagnostic studies. It also offers enhanced spatial integration that resulting in better contouring and targeting of prostate lesions.

In the light of current issues, the next question is whether PSMA PET imaging could add to the detection of prostate cancer. Several retrospective case-report studies reported promising results regarding the improved diagnostic accuracy of prostatic PSMA PET/CT . Recently, in the PRIMARY trial, 291 men received successively MRI, PSMA PET/CT and systematic ± MRI-targeted biopsies. Despite similar PPV between imaging methods, the main advantage of PSMA was in men with equivocal MRI. Indeed, they found that 90% of csPCa was identified by PSMA PET/CT in this subgroup and paved the way for further investigation. This finding was confirmed in the most recent systematic review and meta-analysis.

The aim of this prospective study is to evaluate the added-value of PSMA PET in detecting prostate cancer in patients who are candidates for biopsy with equivocal MRI.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria for inclusion in the study:

* Men ≥ 18 years of age
* Multiparametric MRI within the previous 6 months
* At least one lesion PI-RADS 3
* Able to provide written informed consent

Exclusion Criteria:

Eligible subjects must not meet any of the exclusion criteria listed below:

* Previous prostate cancer diagnostic on MRI-targeted biopsy
* At least one lesion PI-RADS 4-5
* Negative MRI (PI-RADS 1-2)
* Previous treatment for prostate cancer 11
* Contraindication to PSMA PET and/or MRI and/or prostate biopsy
* Low quality of MRI defined by a PI-QUAL score of 1 or 2
* Any medical condition that may interfere with the study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men ≥ 18 years of age
Enrollment: 68 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with clinically significant prostate cancer detected by PSMA PET-targeted biopsy | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium